CLINICAL TRIAL: NCT01983293
Title: Cardiac Resynchronization Therapy (CRT) Implant Strategy Using the Longest Electrical Delay for Non-left Bundle Branch Block Patients (ENHANCE CRT). A Prospective, Randomized, Postmarket, Pilot Study.
Brief Title: CRT Implant Strategy Using the Longest Electrical Delay for Non-left Bundle Branch Block Patients
Acronym: ENHANCE CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60037834
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Non-left Bundle Branch Block; Ischemic or Non-ischemic Cardiomyopathy
Keywords: Non-left bundle branch block; QLV; LV lead pacing location; CRT-D
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- QLV based implant strategy (Experimental): QLV represents the pacing site with the largest amount of dyssynchrony as measured by the left ventricular electrical delay. The QLV based implant strategy finds the left ventricle vein branch and left ventricular lead cathode with the longest QLV measurement and places the lead at this location and programs the device using this lead cathode.
  Interventions: Device: QLV based implant strategy
- Standard of care implant strategy (Placebo Comparator): The placement of LV lead will be carried out according to the physician's standard of care implant approach.
  Interventions: Device: Standard of care implant strategy

INTERVENTIONS:
Device: QLV based implant strategy
  Arms: QLV based implant strategy
Device: Standard of care implant strategy
  Arms: Standard of care implant strategy

SUMMARY:
The purpose of this study is to analyze the effect of left ventricular lead pacing location in the non-left bundle branch block (non-LBBB) heart failure patient population. The left ventricular lead pacing location will be guided by either the pacing site with the largest amount of dyssynchrony as measured by the LV electrical delay (QLV) or the physician's standard of care implant approach.

DETAILED DESCRIPTION:
This is a prospective, pilot, multi-center, double-blinded, randomized post-market study to assess the effect of left ventricular lead pacing location (guided via QLV measurement vs. standard of care approach) in non-LBBB patients.

In the QLV arm the physician will:

1. Assess two branches of the coronary sinus - a non-traditional vessel (inclusive of the anterior region) will be tested first and a traditional free lateral branch will be tested second for LV lead placement.
2. Measure QLV for each of the four cathodes of the left ventricular lead in each branch.
3. Choose the vein branch and cathode with the longest QLV measurement and program a vector based on that cathode.

In the standard of care group, the left ventricular lead placement will be carried out according to the physician's standard of care implant approach.

The impact of the left ventricular lead position will be evaluated based on the patient's response to CRT utilizing the Clinical Composite Score (cardiovascular death, heart failure hospitalizations, New York Heart Association (NYHA) class, and Patient Global Assessment). Authorized site personnel conducting the NYHA class assessment and Patient Global Assessment will be blinded to the randomization assignment and lead implant technique.

ELIGIBILITY:
Inclusion Criteria:

* Have non-LBBB morphology (includes complete right bundle branch block and intraventricular conduction delay with a QRS duration ≥ 120ms)
* Have the following indication per the 2013 updated American College of Cardiology Foundation/American Heart Association/Heart Rhythm Society guidelines:

  * Left ventricular ejection fraction (LVEF) ≤ 35%, sinus rhythm, ischemic or non-ischemic cardiomyopathy, a non-LBBB pattern with QRS duration ≥ 120 ms, and NYHA) class III/ambulatory class IV on guideline directed medical therapy
* Receiving a new CRT implant or undergoing an upgrade from an existing implantable cardioverter defibrillator or pacemaker implant with no more than 10% right ventricular pacing
* Are 18 years or older, or of legal age to give informed consent specific to state and local law
* Ability to provide informed consent for study participation and is willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Irreversible occlusion of venous access that will prevent placement of the CRT system either through the right or left upper extremity venous system
* Undergoing left ventricular lead placement via a surgical or epicardial approach
* Cardiomyopathy due solely to valvular disease that is not repaired/replaced
* Enrolled or intend to participate in a clinical drug and/or device study, which could confound the results of this trial as determined by St. Jude Medical, during the course of this clinical study
* LBBB: QRS width ≥ 120 ms, with predominantly negative QRS in lead V1, and upright, monophasic QRS in leads I and V6
* Incomplete right bundle branch block - intraventricular conduction delay with a QRS duration between 110 and 119ms
* Persistent or permanent atrial fibrillation
* Pacemaker dependent
* Patients who are being upgraded primarily due to right ventricular pacing
* Women who are pregnant or who plan to become pregnant during the clinical trial
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2013-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet Singh, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (32):
- United States (32):
  - Glendale Adventist Medical Center, Glendale, California
  - USC University Hospital, Los Angeles, California
  - Mission Hospital, Mission Viejo, California
  - St. Joseph's Medical Center, Stockton, California
  - Baker-Gilmour Cardiovascular Institute, Jacksonville, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Heart Associates - Riverdale, Riverdale, Georgia
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Oschner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - United Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Northshore University Hospital, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Ohio State University, Columbus, Ohio
  - Sutherland Cardiology Clinic, Germantown, Tennessee
  - Cardiovascular Associates, PC, Kingsport, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Baylor Regional Center at Plano, Plano, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Cardiovascular Associates of Virginia, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh JP, Berger RD, Doshi RN, Lloyd M, Moore D, Daoud EG; ENHANCE CRT Study Group. Rationale and design for ENHANCE CRT: QLV implant strategy for non-left bundle branch block patients. ESC Heart Fail. 2018 Dec;5(6):1184-1190. doi: 10.1002/ehf2.12340. Epub 2018 Sep 27. PMID 30264456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 248 subjects, with 247 having an attempted implant. Of the 247 subjects with an attempted implant, three subjects were excluded from analysis based on having a LBBB morphology and two excluded based on QRS duration <120 ms.
Groups:
- QLV Study Arm: The QLV study arm includes those patients randomized to receive the placement of the left ventricular CRT lead based on the site of latest electrical delay within the left ventricle.
- Standard of Care Study Arm: The Standard of Care study arm includes those patients randomized to receive the placement of the left ventricular CRT lead based on the investigator's standard of care implant approach.
Period: Overall Study
Arm/Group | QLV Study Arm | Standard of Care Study Arm
Started | 161 | 81
Completed | 128 | 62
Not Completed | 33 | 19
Not completed — Withdrawal by Subject | 29 | 15
Not completed — Missing 12-month visit | 3 | 3
Not completed — Missing NYHA/Patient Global Assessment | 1 | 1

BASELINE CHARACTERISTICS:
Population: The study enrolled 248 subjects, with 247 having an attempted implant. Of the 247 subjects with an attempted implant, three subjects presented with a LBBB morphology and two with QRS durations <120 ms. Therefore, a total of 242 subjects are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | QLV Study Arm | Standard of Care Study Arm | Total
Number analyzed (Participants) | 161 | 81 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study enrolled 248 subjects, 247 having an attempted implant. Three subjects presented with a LBBB morphology and two with QRS durations <120 ms.
  years | 65.7 (12.1) | 64.1 (13.3) | 65.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study enrolled 248 subjects, 247 having an attempted implant. Three subjects presented with a LBBB morphology and two with QRS durations <120 ms.
  Participants
    Female | 27 | 21 | 48
    Male | 134 | 60 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 17
  Not Hispanic or Latino | 147 | 75 | 222
  Unknown or Not Reported | 2 | 1 | 3
NYHA Classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) functional classification has 4 categories:
  Class I (least severe) : No limitation of physical activity Class II: Slight limitation of physical activity Class III: Marked limitation of physical activity Class IV (most severe): Unable to carry on any physical activity without discomfort
  Participants
    NYHA II | 0 | 1 | 1
    NYHA III | 157 | 71 | 228
    NYHA IV | 4 | 9 | 13
Type of Cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic | 100 | 45 | 145
  Non-ischemic | 55 | 33 | 88
  None | 6 | 3 | 9
Types of QRS Morphology [Count of Participants; unit: Participants] — Type of QRS complex morphology was assessed by investigators based on 12-lead ECGs acquired.The QRS complex is typically the main spike seen on an ECG and represents the depolarization of the ventricles of the heart. Main criteria used to assess morphology are athe width and height of the QS complex along with certain patterns.
  Participants
    Intraventricular Conduction Delay | 55 | 33 | 88
    Right Bundle Branch Block | 86 | 36 | 122
    Right Bundle Branch/Left Anterior Fascicular Block | 15 | 9 | 24
    Right Bundle/Left Posterior Fascicular Block | 2 | 1 | 3
    Other | 3 | 2 | 5
QRS Duration [Count of Participants; unit: Participants] — QRS duration is the width of the QRS complex usually measured in milliseconds.
  Participants
    120-149 msec | 75 | 33 | 108
    >= 150 msec | 86 | 48 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improved Clinical Composite Score
Description: Evaluate the Clinical Composite Score (CCS) at 12 months in NLBBB patients using a standard of care vs. latest electrical delay (QLV) implant strategy. The CCS has 4 components: New York Heart Association (NYHA) functional classification, Patient Global Assessment (PGA), heart failure (HF) events, cardiovascular death. NYHA Class ranges from Class I (least severe) to Class IV (most severe); possible PGA responses are "markedly worse", "moderately worse", "slightly worse", "no change", "slightly better", "moderately better, "markedly better". CCS components were used to classify or score subjects as "IMPROVED" (at least one-class improvement in NYHA Class or improvement by PGA "moderately" or "markedly" better AND no HF events AND no cardiovascular death), or "WORSENED" (worsening in NYHA Class OR worsening by PGA "moderately" or "markedly" worse OR presence of HF events OR Cardiovascular death, or "UNCHANGED" (neither "improved" or "worsened"). Note CCS is not a numeric score.
Time Frame: 12 months
Population: Of the 242 subjects enrolled, 44 withdrew for reasons other than cardiac death, six had a missing 12-month visit for reasons other than a heart failure event and two had missing Patient Global Assessments or NYHA classification assessments. As a result, the primary endpoint analysis included 190 enrolled subjects (128 QLV arm; 62 control arm).
Measure: Count of Participants; unit: Participants
Arm/Group | QLV Study Arm | Standard of Care Study Arm
Number analyzed (Participants) | 128 | 62
Participants | 86 | 45
Statistical Analysis 1: Comparison: QLV Study Arm vs Standard of Care Study Arm; Test type: Superiority; p = 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a time period of 1 year from enrollment
Description: Adverse events are any unfavorable clinical event which impacts, or has the potential to impact the health or safety of a patient caused by or associated with a study device or intervention. Adverse events are classified as complication or observations.
  Complications: Adverse events that require invasive intervention.
  Observations: Adverse events that can be managed without invasive intervention.
Groups:
- Standard of Care: In the control arm, investigators implanted the LV lead without the use of QLV measurements and instead used standard practices to identify the most suitable LV lead location
- QLV Based Lead Implant: In the QLV arm, the implanting physician assessed the QLV in at least two main branches of the coronary sinus for LV lead placement
Arm/Group | Standard of Care | QLV Based Lead Implant
All-Cause Mortality (participants affected / at risk) | 4/62 | 9/128
Serious Adverse Events (participants affected / at risk) | 4/62 | 8/128
Other Adverse Events (participants affected / at risk) | 14/62 | 31/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=62) | QLV Based Lead Implant (N=128)
Bleeding/Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lead Dislodgement Or Migration (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial Or Ventricular Arrhythmia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lead Fracture (Product Issues) | 0 (0) | 1 (1)
Therapy For Non-Ventricular Rhythm (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=62) | QLV Based Lead Implant (N=128)
Atrial Or Ventricular Arrhythmia (Cardiac disorders) | 1 (3) | 5 (5)
Bleeding/Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Elevated Pacing Thresholds (Product Issues) | 1 (1) | 4 (5)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Local Tissue Reaction; Formation Of Fibrotic Tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Loss Of Capture (Product Issues) | 1 (1) | 2 (2)
Oversensing (Product Issues) | 2 (2) | 3 (3)
Phrenic Nerve/Diaphragmatic Stimulation (Product Issues) | 3 (4) | 5 (6)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rise In Threshold And Exit Block (Product Issues) | 1 (1) | 2 (2)
Undersensing (Product Issues) | 1 (1) | 2 (2)
Other: Back Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Decompensated Systolic Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Other: Desaturation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Device Insertion Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Device Insertion Site Pain (Intermittent) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Device Reset To Back Up Vvi (Product Issues) | 0 (0) | 1 (1)
Other: Device Site Burning (Intermittent) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Device Site Numbness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Device Site Pain (Injury, poisoning and procedural complications) | 3 (3) | 8 (8)
Other: Device Site Redness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other: Diaphragm Stimulation While Lying Supine (Product Issues) | 0 (0) | 1 (1)
Other: Dysphagia (General disorders) | 0 (0) | 1 (1)
Other: Dysphagia And Dysguesia (General disorders) | 1 (1) | 0 (0)
Other: Elevated Lv Capture Threshold (Product Issues) | 0 (0) | 1 (1)
Other: Itching (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Left Clavicle Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Left Shoulder Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Left Shoulder Pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Other: Left Upper Extremity Edema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Other: Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Other: Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other: Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Worsening Heart Failure Due To Crt (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT01983293/Prot_SAP_ICF_001.pdf